CLINICAL TRIAL: NCT04684433
Title: Surgery in the Time of COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Pierre Wauthy, Medical Director, Brugmann University Hospital
Other Study IDs: CHUB-Farid
Record Dates: First submitted 2020-12-23; First posted 2020-12-24 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical intervention: Patients who had a surgical procedure since the start of the lockdown in Belgium due to the COVID19 pandemic (16 of March 2020 to the 12 of April 2020.
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
The ongoing coronavirus disease 2019 (COVID-19) which started in China, was declared on the 11th of March as a global pandemic 2020 by the World Health Organization (WHO).

Governments around the world have introduced differing forms of lock downs since the start of the pandemic demanding citizens to confine to their homes and go out only in necessity to minimize exposure to the virus. The response was observed in the emergency departments and the number of patients who presented for non-Covid issues drastically reduced.

Hospitals activated their mass casualty management plans and have reorganized and overstretched their capacity to be able to absorb both the influx of patients with the virus and those with other conditions.

Part of that reorganization was reducing the surgical activity. The main focus was shifted to patients who are considered urgent and elective surgery were postponed. Hence only surgical emergencies were maintained. Many did not present to the emergency department for fear to contract the virus and from a sense of national and global solidarity against that pandemic.

Whereas these measures are essential to prevent the spread of the virus, it may be hypothesized that for non-Covid issues, including surgical emergencies, patients may present late to the emergency department due to fear of contracting the infection in hospital. This would delay their management and lead to a worsened symptomology on presentation requiring a more complex surgical intervention with an increased complication profile.

The investigators present initial data from four major hospitals in Belgium, characterizing surgical emergencies that were managed since the start of the pandemic and discuss the repercussion the pandemic has on management of urgent surgical patients and most likely evolution of surgery after the pandemic.

ELIGIBILITY:
Inclusion Criteria:

Patients who had a surgical procedure since the start of the lock down in Belgium due to the COVID19 pandemic (16 of March 2020 to the 12 of April 2020).

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patient that have benefited of a surgical intervention since the start of the COVID19 pandemic in Belgium and specifically the 16 th of March 2020 (lock down) to 12 of april 2020. The involved hospitals are: Brugmann hospital, UZ Brussel Hospital, Erasme Hospital and Saint Pierre Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 707 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Surgery code | 5 minutes
  Type of surgery as defined by the surgery code
Urgency | 5 minutes
  Degree of urgency of the surgery
Type of anesthesia | 5 minutes
  Type of anesthesia
Delay between surgery and first symptoms | 5 minutes
  Delay between surgery and first symptoms
Surgery duration | 5 minutes
  Surgery duration (anesthesia included)
Hospital stay (in days) | 5 minutes
  Hospital stay (in days)
Intensive care unit stay (in days) | 5 minutes
  Intensive care unit stay (in days)
Post-op complications | 5 minutes
  Post-op complications
Covid status before surgery | 5 minutes
  Covid status before surgery (positive=1, negative=0 )
Covid status post-surgery | 5 minutes
  Covid status post-op (positive=1, negative=0 )
COVID19 Diagnosis by CT scan | 5 minutes
  COVID19 Diagnosis confirmed by CT scan of the thorax (Yes=1, No=0)
COVID19 Diagnosis by swab test | 5 minutes
  COVID19 Diagnosis by swab test (Yes=1, No=0)
COVID 19 Diagnosis by antibody test | 5 minutes
  COVID 19 Diagnosis by antibody test (Yes=1, No=0)
COVID19 symptoms - dry cough | 5 minutes
  dry cough (Yes=1, No=0)
COVID19 symptoms - fever | 5 minutes
  fever (Yes=1, No=0)
COVID19 symptoms - myalgia | 5 minutes
  myalgia (Yes=1, No=0)
COVID19 symptoms - anosmia | 5 minutes
  anosmia (Yes=1, No=0)
COVID19 symptoms -respiratory distress | 5 minutes
  respiratory distress (Yes=1, No=0)
Treatment for COVID19 - Plaquenil | 5 minutes
  Plaquenil (Yes=1, No=0)
Treatment for COVID19 - Antivirals | 5 minutes
  Antivirals (Yes=1, No=0)
Need for intubation | 5 minutes
  Need for intubation (Yes=1, No=0)
Death | 5 minutes
  Mortality (Yes=1, No=0)

SECONDARY OUTCOMES:
Age | 5 minutes
  Patient age
Gender | 5 minutes
  Patient gender
Ethnicity | 5 minutes
  Patient ethnicity
BMI | 5 minutes
  Patient Body Mass Index
Comorbidities | 5 minutes
  Patient comorbidities

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Farid, Study Director — CHU Brugmann
Locations (4):
- Belgium (4):
  - St Pierre, Brussels
  - CHU Brugmann, Brussels
  - Erasme, Brussels
  - UZ Brussel, Brussels

IPD SHARING:
Plan to Share IPD: No